CLINICAL TRIAL: NCT04520529
Title: Identification of Prognostic Factors and New Therapeutic Targets in Cutaneous Lymphomas
Acronym: LYMPHOTEQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP190179
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Cutaneous Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with primary cutaneous lymphoma (Other)
  Interventions: Other: Biologic Samples

INTERVENTIONS:
Other: Biologic Samples — * An additional punch from lesion skin as part of a skin biopsy performed as part of routine care.
  * an additional blood sample will be collected for research during a blood test performed as part of the patient's routine care.
  * In patients with clinical superficial lymphadenopathy or detected by imaging, and undergoing a superficial lymph node biopsy as part of the care, a core biopsy will be dedicated to research.

SUMMARY:
Cutaneous lymphomas are a heterogeneous group of extra-nodal lymphomas. The prognosis of cutaneous lymphomas is extremely variable from one subject to another. In the majority of cases, there is no cure for cutaneous lymphomas. Cutaneous lymphomas primarily affect the skin, and secondarily the blood, lymph nodes and possibly other organs. The discovery of new molecular prognostic factors will allow a better identification of patients at high risk of aggressive evolution and the implementation of a personalized therapeutic strategy. The identification of new therapeutic targets is necessary in order to develop new innovative treatments for cutaneous lymphomas.The primary objective is to identify novel molecular prognostic factors associated with 5-year overall survival in cutaneous lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Informed consent signed by the patient
* Suspicion of primary cutaneous lymphoma or confirmed lymphoma according to WHO/ISCL/EORTC criteria

Exclusion Criteria:

* Patient under guardianship or curatorship
* Lack of affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2045-09-30 (Estimated); Study Completion 2050-09-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
Progression free survival | 5 years
Progression free survival | 10 years
Overall survival | 10 years

IPD SHARING:
Plan to Share IPD: Undecided